CLINICAL TRIAL: NCT05373888
Title: Prospective, Non-interventional, Post-Market Clinical Follow-up Investigation of the Safety and Performance of Flexima®/Softima® Stoma Appliances in Enterostomy Patients
Brief Title: Safety and Performance of Flexima®/Softima® Stoma Appliances in Enterostomy Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: BBraun Medical SAS (Industry)
Responsible Party: Sponsor
Other Study IDs: OPM-O-H-2005
Record Dates: First submitted 2022-05-10; First posted 2022-05-13 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Enterostomy; Stoma Ileostomy; Stoma Colostomy
Keywords: enterostomy; colostomy; ileostomy; stoma; jejunostomy; stoma appliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Main: Enterostomy patients, including colostomates, ileostomates or jejunostomates.
  Interventions: Device: Flexima®/Softima® stoma bags

INTERVENTIONS:
Device: Flexima®/Softima® stoma bags — One piece stoma bags for enterostomates available as:
  * Closed (flat and convex)
  * Drainable with Roll'Up (flat and convex)
  * High flow with tape outlet (flat)

SUMMARY:
The study is designed as a non-interventional, prospective, international, multi-center, post market follow-up investigation. The product under investigation will be used in routine clinical practice and according to Instructions for Use (IFU). The data obtained during routine clinical use will be documented in electronic Case Report Forms (eCRF).

The investigation will consist of an enrolment visit (Visit 1, or V1) and a final visit (Visit 2, or V2). The duration between the two visits is 14 (±3) days.

DETAILED DESCRIPTION:
Details of the procedures performed at each visit follow.

#A ENROLMENT VISIT (Visit 1, onsite)

The following procedures will be performed:

* Informed consent
* Eligibility assessment
* Record demographics
* Record medical and surgical history (including stoma details)
* Record details of the appliance currently used, which could be different than a Flexima®/Softima®. However, participation in the investigation requires a Flexima®/Softima® appliance be used.
* Peristomal skin assessment (DET scoring)
* Discuss investigation requirements with the participant, including the need of adequately completing the patient's diary
* Start recording adverse events and concomitant medications

  * B 14 (±3 DAY) DEVICE WEARING TIME (telephone follow-up)

During the wearing time, the following procedures will be done:

* The clinical site personnel will follow-up with the participants by telephone as required
* Participants will complete the patient's diary, which includes a record of appliance changes and assessment of leakages
* Record adverse events and concomitant medications (via telephone follow-up)

  * C FINAL VISIT (Visit 2, onsite)

During the final visit, the following procedures will be done:

* Peristomal skin assessment (DET scoring)
* Participant evaluation of device performance (see 8.2.7)
* The responsible site personnel will review the patient's diary together with the patient. Any missing data will be discussed with the patient and, if possible, completed. In case it can't be completed, clarification notes explaining the reason for the missing data are to be added to the patient's diary (e.g. details forgotten)
* Record adverse events and concomitant medications

ELIGIBILITY:
Inclusion Criteria:

* Patients for whom the use of a Flexima®/Softima® appliance is indicated and has been decided within the regular planning of their treatment. Both, new users or users already using Flexima®/Softima® appliances are eligible for participation.

Exclusion Criteria:

* Patients under 18 years old
* Patients who are mentally or linguistically unable to understand the aim of the investigation; or unable to comply with the investigation procedures.
* Patients taking part in another clinical investigation which could have an impact on the current investigation.
* Patient vulnerable. Vulnerable patients are adults unable to express their consent, patients under legal protection, patients deprived of their liberty by a judicial or administrative decision, patients subject to psychiatric care against their will and pregnant, parturient or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Enterostomy patients, including colostomates, ileostomates or jejunostomates.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with at least one adverse device effect (ADE) as judged by the clinician. | 14 days
  The primary variable is the number of patients with at least one adverse device effect (ADE) as judged by the clinician.
  The occurrence of any of the following events in the peristomal skin may be considered related to the use of the stoma appliance (ie, ADEs):
  * Allergic contact dermatitis
  * Mechanical dermatitis - trauma
  * Irritant-chemical dermatitis
  * Infectious conditions
  * Any other appliance related complication (as judged by the clinician)

CONTACTS AND LOCATIONS:
Locations (1):
- Fundacion Jimenez Diaz, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided